CLINICAL TRIAL: NCT05105815
Title: An Exploratory Study on the Safety and Effectiveness of Autoimmune Cell Therapy Sensitized With Liver Cancer Neoantigen in Patients With High Risk of Recurrence After Surgical Resection of Primary Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Autoimmune Cell Therapy for Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Beijing Immupeutics Medicine Technology Limited (Industry); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Zhang, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-567
Record Dates: First submitted 2021-10-23; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPM001 (Experimental): A neoantigen/tumor-specific antigen sensitized autoimmune cell injection
  Interventions: Biological: IPM001

INTERVENTIONS:
Biological: IPM001 — IPM001 will be used against tumor cells

SUMMARY:
In this study, safety and effects of IPM001 vaccine on human hepatocellular carcinoma are going to be investigated, IPM001 is a neoantigen/tumor-specific antigen sensitized autoimmune cell injection

ELIGIBILITY:
Inclusion Criteria:

* understand and voluntarily sign a written informed consent;
* Age: from 18 to 75 years, No restriction on gender;
* Patients must have primary hepatocellular carcinoma;
* Clinical stage: stage Ia~III a;
* Child-pugh score ≤7;
* HLA-A02 and consistent with ≥1 NeoAg or ≥2 aeTSA peptide bank;
* ECOG PS score: 0~2;
* Laboratory values as follow:
* White blood cell count ≥ 3×109/L; Neutrophils: more than 1.5 × 109/L; Hemoglobin: more than 85g/L; Platelets: more than 5 × 1010/L; Total bilirubin:≤2 × ULN; Serum AST(GOT) and ALT(GPT)≤2.5 × ULN; Albumin ≥3.0 g/dL (30 g/L); Serum creatinine: less than 1.5 × ULN; Coagulation time was basically normal, PT extension ≤4s; No serious cardiopulmonary disease;
* Blood collection body weight: male > 50 kg, female > 45 kg;
* No obvious hereditary diseases;
* Expected survival: more than 6 months;

Exclusion Criteria:

* Patient has known distant organ metastasis;
* Suffer from lymphoma or leukemia or MDS (myelodysplastic syndrome), etc.;
* Woman be pregnant or lactating;
* Suffer from mental or neurological diseases that are resistant to control;
* The investigator judges that it is not suitable to participate in this clinical research (such as poor compliance, etc.);
* Patients infected with human immunodeficiency virus (commonly known as AIDS) or Treponema pallidum (commonly known as syphilis);
* Patients with a history of other malignant tumors in the past 5 years;
* Organ transplantation or Myelosuppression;
* History of drug abuse or alcohol abuse;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 18 months
  The time between the NeoAg/aeTSA CTL initiation and the onset of tumor recurrence or death from any cause

SECONDARY OUTCOMES:
OS | 24 months
  From the beginning of NeoAg/aeTSA CTL initiation to the time of death from any cause
EORTC-QLQ30 | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No